CLINICAL TRIAL: NCT06988488
Title: A Phase 1b/2a, Multicenter, Open-label Study to Determine the Recommended Dose and Schedule, and Evaluate the Safety and Preliminary Efficacy of Mezigdomide in Combination With Elranatamab in Participants With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study to Determine the Recommended Dose and Schedule, and Evaluate the Safety and Preliminary Efficacy of Mezigdomide in Combination With Elranatamab in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA057-1040; 2025-522090-11 (Other: EU CTR); U1111-1317-4901 (Other: WHO)
Expanded Access: NCT06994117 (Available)
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental)
  Interventions: Drug: Elranatamab; Drug: Mezigdomide; Drug: Dexamethasone
- Phase 2 (Experimental)
  Interventions: Drug: Elranatamab; Drug: Mezigdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elranatamab — Specified dose on specified days
  Other Names: Elrexfio; PF-0686313
Drug: Mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480
Drug: Dexamethasone — Specified dose on specified days
  Other Names: Decadron®

SUMMARY:
The purpose of this study is to evaluate the preliminary safety and determine the RP2D of mezigdomide in combination with elranatamab in participants with relapsed and refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 with history of relapsed and refractory multiple myeloma (RRMM) treated with 2 to 4 prior lines of anti-myeloma therapy (Phase 1) or 1 to 3 prior lines of anti-myeloma therapy (Phase 2).
* Measurable MM by local laboratory.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1.
* Adherence to contraception requirements.

Exclusion Criteria:

* Prior treatment with mezigdomide.
* Prior treatment with T cell engaging or T cell engager (TCE).
* Prior treatment with B cell-maturation antigen (BCMA)-targeting therapy, with the exception of participants who have received autologous BCMA-targeted CART-cell therapy> 6 months from the start of study therapy
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From first participant first visit until 28 days after the last mezigdomide dose or 90 days after last elranatamab dose, whichever is longer
Number of participants with Serious AEs | From first participant first visit until 28 days after the last mezigdomide dose or 90 days after last elranatamab dose, whichever is longer
Number of participants with AEs meeting protocol-defined DLT criteria | From first participant first visit until 28 days after the last mezigdomide dose or 90 days after last elranatamab dose, whichever is longer
Number of participants with AEs leading to discontinuation | From first participant first visit until 28 days after the last mezigdomide dose or 90 days after last elranatamab dose, whichever is longer
Number of deaths | From first participant first visit until 28 days after the last mezigdomide dose or 90 days after last elranatamab dose, whichever is longer
Recommended Phase 2 Dose (RP2D) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)

SECONDARY OUTCOMES:
International Myeloma Working Group (IMWG) Uniform Response Criteria: Overall Response Rate (ORR) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
IMWG Uniform Response Criteria: Complete Response Rate (CRR) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
IMWG Uniform Response Criteria: Very Good Partial Response Rate (VGPRR) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
IMWG Uniform Response Criteria: Time to Response (TTR) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
IMWG Uniform Response Criteria: Duration of Response (DOR) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
IMWG Uniform Response Criteria: Progression-free Survival (PFS) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
IMWG Uniform Response Criteria: Overall Survival (OS) | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
Number of participants who achieve minimal residual disease (MRD) negativity | From first participant enrollment until the last participant is no longer evaluable for response or has progressed or the last survival follow-up (At approximately 5 years)
  Defined as less than 1 in 10^5 nucleated cells in BMA for participants who achieve CR or better at any time after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale New Haven Hospital-Smilow Cancer Center, New Haven, Connecticut
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Local Institution - 0026, Vancouver, British Columbia
  - Local Institution - 0027, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (2):
  - Local Institution - 0030, Suzhou, Jiangsu
  - Local Institution - 0031, Shanghai, Shanghai Municipality
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
- Greece (2):
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
- Norway (2):
  - St. Olavs Hospital, Trondheim, Sør-Trøndelag
  - Sykehusapoteket Ull, Oslo
- Spain (2):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
- United Kingdom (3):
  - University College London Hospital, London, England
  - Royal Marsden Hospital (Sutton), London, Sutton
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html